CLINICAL TRIAL: NCT01481870
Title: Randomized Comparison of Sequential Therapies With Sunitinib and Sorafenib in Advanced Renal Cell Carcinoma
Brief Title: Comparison of Sequential Therapies With Sunitinib and Sorafenib in Advanced Renal Cell Carcinoma
Acronym: CROSS-J-RCC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yamagata University (Other)
Responsible Party: Principal Investigator, Yoshihiko TOMITA, Clinical Professor, Head of Department of Urology, Yamagata University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CROSS-J-RCC; UMIN000003040 (Other: Japanese University Hospital Medical Informaton Network (UMIN))
Record Dates: First submitted 2011-11-17; First posted 2011-11-30 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: renal cell carcinoma; sorafenib; sunitinib; crossover
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sorafenib-sunitinib (Active Comparator): Sorafenib is first line treatment followed by sunitinib.
  Interventions: Drug: Sorafenib-sunitinib
- Sunitinib-sorafenib (Active Comparator): Sunitinib is first line treatment followed by sorafenib.
  Interventions: Drug: Sunitinib-sorafenib

INTERVENTIONS:
Drug: Sorafenib-sunitinib — sorafenib 400mg b.i.d. followed by sunitinib treatment when progression is observed
  Arms: Sorafenib-sunitinib
Drug: Sunitinib-sorafenib — sunitinib 50mg q.d. 4 weeks on two weeks off followed by sorafenib treatment when progression is observed
  Arms: Sunitinib-sorafenib

SUMMARY:
The clinical benefits of sunitinib and sorafenib have been demonstrated in patients with cytokine-refractory metastatic renal cell carcinoma. Sunitinib has also been shown to improve progression free survival and overall survival in a comparative study with interferon-alpha. When sunitinib is used as first-line molecular-targeted therapy, switching to sorafenib is one of the treatment options after disease progression. Reversely, when sorafenib is used as first-line molecular-targeted therapy, sunitinib is used as second-line therapy. The goal of cancer treatment is cure, and if cure is not possible, it is to prolong survival. In this study, sunitinib or sorafenib will be administered as first-line molecular-targeted therapy and treatment switched to the other test drug, sorafenib or sunitinib, when disease progression is detected to assess which treatment sequence produces longer progression free survival and offers a better safety profile (causing fewer adverse events). The purpose of this trial is to compare progression free survival of first line sunitinib versus sorafenib, and that of two treatment sequences, i.e. sunitinib followed by sorafenib versus sorafenib followed by sunitinib.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-80 years old, both inclusive
* ECOG performance status of 0, 1, or 2
* MSKCC risk of favorable or intermediate
* Histologically confirmed renal cell carcinoma
* No ischemic heart disease
* Laboratory findings meet the following criteria:

  1. Respiratory function: %VC, 80% and FEV1.0,70%
  2. Hematology: white blood cell count4,000/mm3, platelet count100,000/mm3
  3. Clinical chemistry: GOT and GPT within the normal range of each medical institution; total bilirubin <1.5 x ULN
  4. Serum creatinin <2.0mg/dl, blood urea nitrogen (BUN) <25mg/dl
  5. Echocardiographic estimation of left ventricular ejection fraction is higher than the lower limit of reference range of each medical institution.

Exclusion Criteria:

* History of any other malignancy
* Central nervous system metastases. However, patients who remain asymptomatic, have no new or enlarging lesion in the CNS within 6 months of enrollment in this study, and require no corticosteroids may be enrolled.
* History of cardiac infarction, unstable angina, congestive heart failure, or symptomatic peripheral vascular disease within 12 months of enrollment
* History of cerebrovascular disorder including transient ischemic attack (TIA)
* Pregnancy or possible pregnancy at any time during the study
* Ongoing grade 2 adverse event prior treatment
* Prior treatment with any anticancer therapy including cytokine therapy such as interferon-alpha and interleukin-2
* Prior treatment with mTOR inhibitor
* Prior treatment with sunitinib or sorafenib
* Treatment with an test drug in a clinical research within 4 weeks of enrollment in this study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-01; Primary Completion 2013-07 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival in first-line treatment | Time of progression in first line treatment
  From date of randomization until the date of first documented progression of the first line treatment or date of death from any cause, whichever came first, assessed up to 36 months.

SECONDARY OUTCOMES:
Total progression free survival (PFS) in first-line and second-line treatments | Time of progression in second line treatment
  From date of randomization until the date of first documented progression of the second line treatment or date of death from any cause, whichever came first, assessed up to 36 months.

CONTACTS AND LOCATIONS:
Overall Officials: Yoshihiko Tomita, MD, Principal Investigator — Yamagata University Faculty of Medicine
Locations (1):
- Yamagata University Faculty of Medicine, Yamagata, Japan

REFERENCES:
- [Background] Tomita Y, Shinohara N, Yuasa T, Fujimoto H, Niwakawa M, Mugiya S, Miki T, Uemura H, Nonomura N, Takahashi M, Hasegawa Y, Agata N, Houk B, Naito S, Akaza H. Overall survival and updated results from a phase II study of sunitinib in Japanese patients with metastatic renal cell carcinoma. Jpn J Clin Oncol. 2010 Dec;40(12):1166-72. doi: 10.1093/jjco/hyq146. Epub 2010 Aug 16. PMID 20713418
- [Derived] Aldin A, Besiroglu B, Adams A, Monsef I, Piechotta V, Tomlinson E, Hornbach C, Dressen N, Goldkuhle M, Maisch P, Dahm P, Heidenreich A, Skoetz N. First-line therapy for adults with advanced renal cell carcinoma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 May 4;5(5):CD013798. doi: 10.1002/14651858.CD013798.pub2. PMID 37146227
- [Derived] Tomita Y, Naito S, Sassa N, Takahashi A, Kondo T, Koie T, Obara W, Kobayashi Y, Teishima J, Takahashi M, Matsuyama H, Ueda T, Yamaguchi K, Kishida T, Shiroki R, Saika T, Shinohara N, Oya M, Kanayama HO. Sunitinib Versus Sorafenib as Initial Targeted Therapy for mCC-RCC With Favorable/Intermediate Risk: Multicenter Randomized Trial CROSS-J-RCC. Clin Genitourin Cancer. 2020 Aug;18(4):e374-e385. doi: 10.1016/j.clgc.2020.01.001. Epub 2020 Mar 6. PMID 32466961
- See also: UMIN Clinical Trial Registry — https://upload.umin.ac.jp/cgi-open-bin/ctr/ctr.cgi?function=brows&action=brows&type=summary&recptno=R000003325&language=J